CLINICAL TRIAL: NCT01232387
Title: Identification of Early Predictors of Fetomaternal Hemorrhage And Development Of An Automated Screening Strategy For At-Risk Pregnancies
Brief Title: Identification of Early Predictors of Fetomaternal Hemorrhage
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); New York Blood Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0920; KL2RR029885 (NIH)
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Fetomaternal Hemorrhage; Neonatal Anemia
Keywords: Fetomaternal hemorrhage; neonatal anemia; perinatal epidemiology; Kleihauer-Betke; flow cytometry
MeSH Terms: conditions — Fetomaternal Transfusion; Anemia, Neonatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, placenta
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fetomaternal hemorrhage - Mothers: Mothers in Mother-baby pairs in which the testing for fetomaternal hemorrhage on the mother's blood demonstrates the presence of fetal cells.
- Fetomaternal hemorrhage - Babies: Babies in Mother-baby pairs in which the testing for fetomaternal hemorrhage on the mother's blood demonstrates the presence of fetal cells.

SUMMARY:
Objectives: 1) To determine risk factors for fetomaternal hemorrhage. 2) To identify a cost-effective method to detect fetomaternal hemorrhage prior to significant fetal anemia.

Significance/Background: Fetomaternal hemorrhage (FMH) is a condition in which occurs when the placenta transfers blood from the fetus to the mother. Normally, nutrition and gasses pass from mother to baby through the placenta and only waste products pass from baby to mother through the placenta. Whole blood cells do not normally cross the placenta in significant amounts. Mild FMH, where a small amount of whole blood passes from fetus to mother but does not hurt the mother or baby, occurs in about 75% of pregnancies. A pregnant woman does not know this occurs. It is only discovered if a special blood test that is labor-intensive to perform and difficult to interpret called the Kleihauer-Betke acid elution test is done. As mild FMH hurts no one, this test is not part of routine care. In most cases, testing is done only if a baby is born sick with unexplained anemia. Severe FMH, which can cause the baby to become sick from anemia (low red blood cell count) is caused by large blood loss into the mother, occurs in only 1-3 per 1000 births. Severe anemia caused by FMH can result in death of the baby before or after birth, or significant illness in the newborn period. Short term problems for the baby include difficulty breathing, difficulty maintaining blood pressure, and difficulty providing oxygen to all parts of the body. This can cause multiple problems with the function of internal organs including the liver, kidneys, intestines, and brain. Babies who become sick from severe FMH can develop long-term problems including cerebral palsy (a lifelong problem with body movements) and/or mental retardation.

It is not known why some pregnancies are affected by FMH and others are not. It is thought that FMH may occur more frequently now than in the past, but no one knows why. If identified early, FMH is readily treatable by blood transfusion of the baby before or after birth and/or early delivery. Current laboratory testing for FMH is difficult and expensive. There is great need identify high risk patients early in pregnancy in order to treat the condition before the baby gets sick.

Approach: Five hundred women will be asked to participate in the study at the time they are admitted to the Mount Sinai labor floor for delivery at term. After birth, newborns of study mothers will be tested for anemia. Mothers of anemic babies will donate blood for confirmation of FMH by established laboratory methods as well as for development of a new laboratory screening protocol. All mothers will provide medical, social, environmental, and full pregnancy history. Risk factors for FMH will be identified by statistical analysis of this information.

DETAILED DESCRIPTION:
1. Introduction:

   The objective of this study is to identify candidate clinical predictors of fetomaternal hemorrhage (FMH) and to devise a screening strategy to identify pregnancies affected by the condition before the fetus is compromised by severe anemia.

   Fetomaternal hemorrhage is a condition in which the placental barrier fails and the fetus "bleeds" into the maternal circulation. When functioning correctly, the placenta allows transfer of nutrients and waste between the mother and fetus while keeping the cellular components of blood separate. It is not uncommon for small amounts of fetal blood to reach the maternal circulation without adverse effect on the fetus. In fact, mild FMH can be detected in up to 75% of normal pregnancies. In approximately 3 in 1000 pregnancies, however, the volume of fetal blood transferred to the mother causes clinically-significant anemia in the fetus. Fetal anemia can cause significant morbidity and mortality. In fetuses who survive severe anemia, life-long disability is common.

   Diagnosis of FMH is most commonly made after an adverse fetal or neonatal outcome has occurred, indicating the need for testing. Early risk factors for FMH are unknown. Clinical predictors of FMH have been suggested, but have not been born out in retrospective study. Current standard of care testing for FMH, the Kleihauer-Betke (KB) acid elution test, is labor-intensive and time-consuming, and therefore expensive. Additionally, the KB test is observer-dependent and can be significantly affected by variations in sample preparation. No screening protocol for FMH with automated laboratory testing appropriate for use in the general pregnant population exists.

   Specific Aim: To identify an appropriate laboratory protocol for diagnosis of fetomaternal hemorrhage by prospective study and to pilot a study intended to determine early clinical predictors of mild fetomaternal hemorrhage.
2. Background and Significance Fetomaternal hemorrhage occurs when the normal flow of blood within the placenta is disrupted and the cellular components of fetal blood cross into the maternal circulation. A healthy placenta permits transfer of dissolved substances between the mother and fetus while keeping the cellular components of the two circulations separate. It is common for the placental filter to "leak" during normal pregnancies, resulting in transfer of small volumes of fetal whole blood into the maternal bloodstream. Volumes of fetal blood under 1 mL can be detected in up to 75% of pregnancies. This volume of blood loss is thought to be clinically insignificant to the fetus. Severe FMH with a large volume of blood transfer from the fetus to the mother is less common. Although the exact volume of blood transfer needed to classify FMH as "severe" is debated, it is clear that significant acute or chronic hemorrhage leads to adverse perinatal outcome. Estimates of the incidence of severe FMH vary, primarily because no comprehensive epidemiologic studies of the condition exist. Estimates based on screening for Rh alloimmunization in Rho(d) negative women suggest that severe FMH occurs in 1-3 of 1000 pregnancies, , but accounts for almost 14% of otherwise unexplained fetal deaths. Large volume FMH can result in severe fetal anemia. Although fetal anemia can manifest in utero with recognized hydrops fetalis or intrauterine growth restriction, more commonly there are no outward signs of FMH-related severe anemia before stillbirth, fetal distress at delivery, or neonatal critical illness. The immediate sequelae of severe FMH for neonates that survive delivery include devastating illnesses such as persistence of the fetal circulation, hypovolemic shock, and hypoxic-ischemic encephalopathy. Ultimate detrimental outcomes include high rates of mental retardation, cerebral palsy, neurologic devastation, and death. Despite these consequences, and a suspected recent rise in incidence of severe FMH, early predictors of severe FMH remain unknown and no cause of hemorrhage can be identified in over 80% of cases. Maternal or pregnancy risk factors appropriate for early screening or diagnosis of severe FMH in the general pregnant population have not been elucidated. , If identified prior to delivery, fetal anemia from FMH can be successfully managed by intrauterine fetal transfusion and delivery prior to the onset of labor. , Outcomes following treatment of fetal anemia with fetal transfusion, even repeated fetal transfusion, are encouraging. Thus, empirical predictors of FMH would offer immediate promise for improving clinical outcomes. The social and financial cost of both initial intensive care and long-term chronic care for children with cognitive and motor disability resulting from FMH is substantial. There is considerable need for early risk identification and a practical screening strategy to mitigate the human and economic costs of severe FMH.

Validated clinical predictors of FMH include decreased fetal movement, sinusoidal fetal heart rate tracing, and hydrops fetalis. , These markers are not useful for prevention of adverse events stemming from FMH as each signifies established severe fetal anemia. Maternal characteristics purported to increase the risk of FMH include hypertension, placental abruption, substance abuse, and trauma. These were evaluated in retrospective study of stillbirths in a 1999 study. None were significantly associated with FMH. Clinical characteristics with suspected association with FMH were evaluated in a 2004 study of Rho(d)-negative women. Only twin gestation was significantly associated with FMH. It is unknown whether the incidence of FMH in multiple gestations is higher than those in singleton pregnancies. No prospective or retrospective epidemiologic survey of FMH in the general pregnant population has been published. No epidemiologic description over the spectrum (mild, moderate, severe) of FMH exists. No series of placental pathology drawn from cases of FMH has been completed.

Currently, even if at-risk pregnancies worthy of screening are identified prior to devastating outcome, laboratory testing for FMH is not straightforward. The most commonly used laboratory test to detect and quantify the volume of fetal blood in the maternal circulation is the Kleihauer-Betke (KB) acid elution test. The reagents for the KB test are relatively inexpensive, but the test is operator-dependent and labor-intensive making it an unappealing candidate for use in expanded screening. The test is based on the fact that an acid eluent will lyse fragile maternal erythrocytes while fetal hemoglobin stabilizes fetal erythrocytes. Maternal blood is obtained and exposed to the acid eluent. Remaining intact fetal cells are stained and counted. Estimates of maternal and fetal total blood volume are then used to calculate the volume of FMH. The KB test is influenced by sample handling, is technician-dependent, and can be inaccurate if patient blood volumes or blood counts are not similar to standard estimates used. It is hypothesized that using maternal height and weight to estimate maternal blood volume for each individual tested can improve the accuracy of KB testing. This method is not widely practiced and has not been validated in the general pregnant population. Such a "corrected KB" warrants further examination.

An additional test that has been explored to avoid some of the pitfalls of KB testing is evaluation of maternal serum alpha-fetoprotein (AFP) levels. The concentration of fetal-derived AFP in the maternal circulation can be used to estimate volume of FMH. As AFP levels vary during and across pregnancies, however, AFP testing is most useful when multiple levels obtained over the course of pregnancy are compared. The vast majority of pregnant women in the United States undergo AFP testing in the second trimester as part of the "quad" or "triple" screening tests for fetal aneuploidy and neural tube defects. Although theoretically viable, no published reports document the use of this second-trimester AFP baseline level for detecting FMH following additional AFP testing closer to term.

The most accurate measurement of FMH developed to date is achieved with flow cytometry (FC) using antibodies specific to the hemoglobin of fetal cells. Cells must be made permeable chemically to permit exposure of the FC antibody to intracellular hemoglobin prior to analysis. Additionally, FC using monoclonal antibodies to fetal hemoglobin has only been documented to reliably diagnose FMH >0.1% in the general clinical population. This is less sensitive than the KB test when performed under standard clinical conditions. Finally, as currently practiced, FC using antibodies to fetal hemoglobin is time-consuming and expensive. This test is therefore not appropriate for large-scale screening at this time.

No series of placental pathology related to FMH has been published. As FMH is thought to be a disease of placental failure, systematic review of placentas of pregnancies affected by FMH could illuminate the pathogenesis of this type of placental abnormality.

Fetomaternal hemorrhage is an under-studied disease entity with significant associated morbidity and mortality. This study aims to identify early clinical predictors of the disease and to develop an automated screening strategy appropriate for wide-spread use. Standard epidemiologic techniques will be used in combination with adaptation of existing laboratory techniques to fully address this problem.

4. Methods: To address these Specific Aims, we propose (1) to test our automated laboratory testing procedures for FMH and (2) to pilot a protocol using the novel automated laboratory testing procedures to identify neonate-mother pairs affected by FMH for identification of early clinical predictors of FMH. This is a pilot prospective nested case-control study.

In collaboration with the Red Cell Physiology laboratory at the New York Blood Center, we have developed a prototype automated assay for FMH using flow cytometry facilities and reagents available at the New York Blood Center.

A convenience sample of women admitted to the Mount Sinai Medical Center labor floor will be selected for this pilot study. Eligible women will be those admitted for term delivery (delivery between 37 0/7 and 41 6/7 weeks from the last menstrual period). Mothers carrying fetuses with known fetal anomaly will be excluded. Women with pre-eclampsia or anomaly of placental implantation (accreta, abruption) will be included, as these conditions may place the pregnancy at risk for FMH but do not currently indicate pregnancy surveillance for fetal anemia. Multiple gestations will be included. Women unable to complete the consent process due to likely precipitous delivery, severe labor discomfort, or fetal distress requiring immediate obstetric intervention will be excluded. Each woman will be enrolled in the study prior to the required antepartum blood draw and/or IV placement, such that a study blood specimen can be obtained with clinically indicated phlebotomy. Study specimens will be banked for batch testing those from pregnancies of interest.

Not all women who donate blood as part of this study will have their blood tested for signs of FMH. Although 5mL of blood will be drawn from eligible consenting women prior to delivery, only specimens of those selected for our stratified sample population based on neonatal hematocrit (HCT) will be tested. All maternal blood drawn will be fixed and/or frozen immediately after phlebotomy for later batched analysis.

Eligible neonates of consenting mothers will have 0.5mL (approximately 3 drops) of blood collected for determination of hematocrit at the time of the required blood draw for the New York State Newborn Screening Program on day two of life. Eligibility will be determined by the absence of a clinical history other than FMH to explain neonatal anemia. Clinical indicators of anemia unrelated to FMH that will be treated as exclusion criteria include hemolytic disease (due to known Rh, Kell, etc sensitization, or Coombs test positive), known significant cord compression at the time of delivery (prolapsed cord, tight cord around the neck or body), twin-to-twin transfusion syndrome recognized as anemia in the donor twin and polycythemia in the recipient twin, and known neonatal blood loss (unclamped cord, laceration). Neonates who have hematocrit measured within the first 48 hours of life for a clinical indication will not have additional blood drawn for this study; results of clinically-indicated samples will be used. All newborns of enrolled mothers will have HCT tested. All mother-baby pairs with demonstrated neonatal anemia (HCT ≤ 50%) will be included in the pilot cohort. In the case of multiple gestation, all siblings will be included for analysis if any demonstrate anemia. Twenty-five percent of neonates with HCT over 50% will also be included in the pilot cohort (every fourth study subject with HCT > 50%). This sampling strategy will allow evaluation over the spectrum of newborn blood counts, over-representing those with anemia.

Maternal blood of study cohort subjects undergo multiple tests for FMH including FC, AFP, and KB. Flow cytometry will be performed at the New York Blood Center. Determination of AFP level and KB testing will be performed by the Mount Sinai Hospital laboratory.

Maternal blood samples will be appropriately fixed at the time of collection, then frozen and batch tested weekly. Any clinically-indicated testing for FMH will be performed independently on blood specimens obtained post-partum, and will not be included in our analysis. All available first trimester AFP testing results will be obtained for cohort mothers. Anthropometric data will be gathered to correct testing results for estimated maternal blood volume based on maternal height and weight. Accuracy of various testing methods at predicting volume of fetal blood in the maternal circulation will be determined by comparison with the KB specimens corrected for actual rather than estimated maternal blood volume.

All placentas of study subjects will be fixed and held by the pathology laboratory for standard one-week duration post-partum. Thirty pregnancies chosen by stratified sampling based on severity of FMH will have the pregnancy placenta(s) subjected to a full pathologic exam. Standard examination techniques including gross and microscopic exam will be used.

After study cohort mothers have been identified, we will collect medical, social, environmental, and full pregnancy history via directed interview. Elements of particular interest will include those hypothesized in the literature to be associated with FMH. Factors suspected in the literature as being associated with FMH include maternal hypertension during pregnancy, maternal pre-eclampsia, maternal trauma during pregnancy, placental abruption, and multiple gestation. The survey tool will investigate these elements of the maternal history as well as take a broad survey of the environmental and social history in an attempt to identify unrecognized clinical predictors of FMH. Maternal subjects will be interviewed during the post-partum stay in the hospital. Data will be used for identification of early risk factors of FMH.

Risk factors will be identified through logistic regression modeling with a multilevel outcome in which FMH is coded as absent (referent), mild, or severe, generating separate odds ratios for mild and severe FMH. The alternate laboratory approaches to identification of FMH will be compared by examining agreement using a kappa statistic, and quantifying agreement across categories.

ELIGIBILITY:
Inclusion Criteria:

* Women admitted for term delivery (delivery between 37 0/7 and 41 6/7 weeks from the last menstrual period) to the Mount Sinai Medical Center

Exclusion Criteria:

* Women carrying fetuses with known fetal anomaly.
* Women unable to complete the consent process due to likely precipitous delivery, severe labor discomfort, or fetal distress requiring immediate intervention.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A convenience sample of women admitted to the Mount Sinai Medical Center labor floor will be selected for this pilot study. Eligible women will be those admitted for term delivery (delivery between 37 0/7 and 41 6/7 weeks from the last menstrual period).
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Neonatal hematocrit | Measured once within the first 72 hours of life
  Blood drawn in conjunction with the mandated New York State Newborn Screening Program specimen

SECONDARY OUTCOMES:
Sign of fetomaternal hemorrhage in maternal blood | Blood drawn once upon admission for labor and delivery.
  Blood drawn in conjunction with clinically indicated antepartum labs

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Stroustrup, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Bowman JM, Pollock JM, Penston LE. Fetomaternal transplacental hemorrhage during pregnancy and after delivery. Vox Sang. 1986;51(2):117-21. doi: 10.1111/j.1423-0410.1986.tb00226.x. PMID 3095989
- [Background] Samadi R, Greenspoon JS, Gviazda I, Settlage RH, Goodwin TM. Massive fetomaternal hemorrhage and fetal death: are they predictable? J Perinatol. 1999 Apr-May;19(3):227-9. doi: 10.1038/sj.jp.7200144. PMID 10685227
- [Background] de Almeida V, Bowman JM. Massive fetomaternal hemorrhage: Manitoba experience. Obstet Gynecol. 1994 Mar;83(3):323-8. PMID 8127519
- [Background] Giacoia GP. Severe fetomaternal hemorrhage: a review. Obstet Gynecol Surv. 1997 Jun;52(6):372-80. doi: 10.1097/00006254-199706000-00022. PMID 9178311
- [Background] Rubod C, Deruelle P, Le Goueff F, Tunez V, Fournier M, Subtil D. Long-term prognosis for infants after massive fetomaternal hemorrhage. Obstet Gynecol. 2007 Aug;110(2 Pt 1):256-60. doi: 10.1097/01.AOG.0000271212.66040.70. PMID 17666598
- [Background] Laube DW, Schauberger CW. Fetomaternal bleeding as a cause for "unexplained" fetal death. Obstet Gynecol. 1982 Nov;60(5):649-51. PMID 7145257
- [Background] Kecskes Z. Large fetomaternal hemorrhage: clinical presentation and outcome. J Matern Fetal Neonatal Med. 2003 Feb;13(2):128-32. doi: 10.1080/jmf.13.2.128.132. PMID 12735414
- [Background] David M, Smidt J, Chen FC, Stein U, Dudenhausen JW. Risk factors for fetal-to-maternal transfusion in Rh D-negative women--results of a prospective study on 942 pregnant women. J Perinat Med. 2004;32(3):254-7. doi: 10.1515/JPM.2004.047. PMID 15188800
- [Background] Fischer RL, Kuhlman K, Grover J, Montgomery O, Wapner RJ. Chronic, massive fetomaternal hemorrhage treated with repeated fetal intravascular transfusions. Am J Obstet Gynecol. 1990 Jan;162(1):203-4. doi: 10.1016/0002-9378(90)90850-7. PMID 2301494
- [Background] Rubod C, Houfflin V, Belot F, Ardiet E, Dufour P, Subtil D, Deruelle P. Successful in utero treatment of chronic and massive fetomaternal hemorrhage with fetal hydrops. Fetal Diagn Ther. 2006;21(5):410-3. doi: 10.1159/000093881. PMID 16912488
- [Background] Brennand J, Cameron A. Fetal anaemia: diagnosis and management. Best Pract Res Clin Obstet Gynaecol. 2008 Feb;22(1):15-29. doi: 10.1016/j.bpobgyn.2007.08.005. Epub 2007 Oct 1. PMID 17904904
- [Background] KLEIHAUER E, BRAUN H, BETKE K. [Demonstration of fetal hemoglobin in erythrocytes of a blood smear]. Klin Wochenschr. 1957 Jun 15;35(12):637-8. doi: 10.1007/BF01481043. No abstract available. German. PMID 13450287
- [Background] Pelikan DM, Scherjon SA, Mesker WE, de Groot-Swings GM, Brouwer-Mandema GG, Tanke HJ, Kanhai HH. Quantification of fetomaternal hemorrhage: a comparative study of the manual and automated microscopic Kleihauer-Betke tests and flow cytometry in clinical samples. Am J Obstet Gynecol. 2004 Aug;191(2):551-7. doi: 10.1016/j.ajog.2004.01.007. PMID 15343236
- [Background] Davis BH, Olsen S, Bigelow NC, Chen JC. Detection of fetal red cells in fetomaternal hemorrhage using a fetal hemoglobin monoclonal antibody by flow cytometry. Transfusion. 1998 Aug;38(8):749-56. doi: 10.1046/j.1537-2995.1998.38898375514.x. PMID 9709783
- [Background] Scholz C, Kachler A, Hermann C, Weissenbacher T, Toth B, Friese K, Kainer F. Flowcytometric assessment of fetomaternal hemorrhage during external cephalic version at term. J Perinat Med. 2009;37(4):334-7. doi: 10.1515/JPM.2009.063. PMID 19290855